CLINICAL TRIAL: NCT05472376
Title: Real-World Outcomes of Anti-VEGF Treatment for Diabetic Macular Edema in Turkey: A Multicenter Retrospective Study, MARMASIA Study Group
Brief Title: Real-Life Study in Diabetic Macular Edema
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Levent Karabas, Prof. Dr., Kocaeli University
Other Study IDs: MARMASIA Study Group
Record Dates: First submitted 2022-07-01; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 3-month follow-up
  Interventions: Other: Retrospective study
- 6-month follow-up
  Interventions: Other: Retrospective study
- 12-month follow-up
  Interventions: Other: Retrospective study
- 24-month follow-up
  Interventions: Other: Retrospective study
- 36-month follow-up
  Interventions: Other: Retrospective study

INTERVENTIONS:
Other: Retrospective study — Retrospective study

SUMMARY:
The goal of this study is to evaluate the real-world outcomes of intravitreal anti-vascular endothelial growth factor (anti-VEGF) treatment in diabetic macular edema (DME) patients.

DETAILED DESCRIPTION:
The study included patients who were being observed in the retina departments of 8 tertiary hospitals in the Northern Marmara Region of Turkey (Istanbul's Asian Side, Kocaeli, and Sakarya). The records of DME patients treated with an anti-VEGF agent between January 2015 and December 2018 were reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic macular edema treated with intravitreal anti-VEGF injection
* Having at least 4 or more annual examination visits

Exclusion Criteria:

* Phacoemulsification surgery in the last 1 month
* PRFK / grid / focal / micropulse in the last 4 months
* Previous intraocular surgery (excluding PPV and phacoemulsification)

Age Groups: Child, Adult, Older Adult
Study Population: The records of DME patients treated with an anti-VEGF agent between January 2015 and December 2018
Sampling Method: Probability Sample
Enrollment: 854 (Actual)
Dates: Start 2020-11-29 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Visit and Intravitreal Injection Numbers | First year
  The primary outcomes were changes in best-corrected visual acuity and central macular thickness in the first year and frequency of visits and intravitreal anti-VEGF injections.

CONTACTS AND LOCATIONS:
Locations (10):
- Turkey (Türkiye) (10):
  - Kocaeli University School of Medicine, Kocaeli, None Selected
  - Marmara University School of Medicine, Istanbul
  - Memorial Şişli Hospital, Istanbul
  - University Health Sciences, Kartal Dr. Lütfi Kırdar Training and Research Hospital, Istanbul
  - University of Health Sciences, Fatih Sultan Mehmet Training and Research Hospital, Istanbul
  - University of Health Sciences, Haydarpaşa Numune Training and Research Hospital, Istanbul
  - University of Health Sciences, Ümraniye Training and Research Hospital, Istanbul
  - University of Health Sciences, Şişli Etfal Training and Research Hospital, Istanbul
  - University of Health Sciences, Derince Training and Research Hospital, Kocaeli
  - Sakarya University School of Medicine, Sakarya

IPD SHARING:
Plan to Share IPD: Undecided